CLINICAL TRIAL: NCT05392348
Title: Regulatory Effect of Stachyose on Gut Microbiota and microRNA Expression in Human
Brief Title: Human Gut Microbiota and microRNA Expression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KY20212094-C-1
Record Dates: First submitted 2021-07-07; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2021-06

CONDITIONS: Gut Microbiota; microRNA
Keywords: stachyose; gut microbiota; microRNA
MeSH Terms: interventions — stachyose; maltodextrin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Control group (Placebo Comparator): Subjects with maltodextrin as intervention，5g/kg·bw/day.
  Interventions: Dietary Supplement: Maltodextrin
- Stachyose intervention group (Experimental): Subjects with stachyose as intervention，5g/kg·bw/day.
  Interventions: Dietary Supplement: stachyose

INTERVENTIONS:
Dietary Supplement: stachyose — Stachyose is a tetrasaccharide consisting of sucrose having an alpha-D-galactosyl-(1->6)-alpha-D-galactosyl moiety attached at the 6-position of the glucose.
  Arms: Stachyose intervention group
Dietary Supplement: Maltodextrin — Maltodextrin is a polysaccharide that is used primarily in foods and beverages as a thickener, sweetener, and/or stabilizer. It is a relatively short-chain polymer (some would call it an oligomer); commercial products contain an average of ≈3 to ≈17 glucose units per chain. It is manufactured by partially hydrolyzing grain starches, usually corn or wheat.
  Arms: Normal Control group

SUMMARY:
In this study, stachyose was used as an intervention factor. We will evaluate changes in fecal gut microbiota and miRNA expression profiles in subjects under stachyose intervention

DETAILED DESCRIPTION:
In the stachyose intervention group, each person in the stachyose intervention group took 5 g of stachyose daily before breakfast, and the administration method was 100 ml of drinking water dissolved and taken orally for two months. Each person in the placebo control group took the same amount of maltodextrin daily. Stool samples of the subjects were collected weekly.

ELIGIBILITY:
Inclusion Criteria:

* healthy human

Exclusion Criteria:

* people who need intake antibiotics，probiotics or its product

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
expression of microRNA | up to 4 weeks
  small rna sequencing valuated the microRNA expression in human
structure of gut microbiota | up to 4 weeks
  16S rDNA sequencing valuated the gut microbiota composition in human

CONTACTS AND LOCATIONS:
Overall Officials: Chao Guo, Study Chair — Xijing Hospital
Locations (1):
- the First Affiliate Hospital of the Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No